CLINICAL TRIAL: NCT03335839
Title: Adjunctive, Low-dose Intracoronary Recombinant Tissue Plasminogen Activator (tPA) Versus Placebo for Primary PCI in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Adjunctive, Low-dose tPA in Primary PCI for STEMI
Acronym: STRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STRIVE.2018
Record Dates: First submitted 2017-11-03; First posted 2017-11-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: tPA
MeSH Terms: conditions — Myocardial Infarction | interventions — Tissue Plasminogen Activator; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intracoronary tPA 10 mg (Experimental)
  Interventions: Drug: tissue plasminogen activator
- Intracoronary tPA 20 mg (Experimental)
  Interventions: Drug: tissue plasminogen activator
- Placebo (Placebo Comparator): saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: tissue plasminogen activator — Recombinant tPA is a fibrin-specific 2nd generation plasminogen activator and thrombolytic drug.
  Arms: Intracoronary tPA 10 mg; Intracoronary tPA 20 mg
Other: Saline — Placebo
  Arms: Placebo

SUMMARY:
STRIVE will evaluate the use of adjunctive, low-dose intracoronary tissue plasminogen activator during primary percutaneous coronary intervention (PCI) for patients with ST elevation myocardial infarction (STEMI) in reducing the incidence of post-procedural myocardial blush (MBG) grade 0/1 or distal embolization.

DETAILED DESCRIPTION:
STRIVE is a prospective, 3-arm, parallel group, blinded, randomized controlled trial evaluating the efficacy of a novel approach to prevent and treat microvascular obstruction thereby reducing major cardiovascular events using intracoronary administration of very low-dose fibrinolytic (tissue plasminogen activator, tPA) directly into the culprit coronary artery during primary PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI undergoing primary PCI and,
2. ECG changes indicating large territory STEMI (defined as ≥2mm ST-segment elevation in 2 contiguous anterior precordial leads; or ≥2mm ST-segment elevation in 2 inferior leads coupled with ST-segment depression in 2 contiguous anterior leads for a total ST-segment deviation of ≥8mm) and,
3. Randomization within 6 to 12 hours of symptom onset and,
4. Large thrombus burden with angiographic TIMI Thrombus Grade ≥3 after guidewire crossing.

Exclusion Criteria:

1. Active internal bleeding or high risk of bleeding or any prior intracranial bleeding.
2. Any other absolute or relative contraindication to fibrinolytic therapy.
3. Administration of a fibrinolytic ≤24hrs prior to randomization.
4. Cardiogenic shock on presentation.
5. Left bundle branch block (excluded because the ECG cannot be evaluated for ST segment resolution, an outcome of the study).
6. Planned upfront use of a glycoprotein IIb/IIIa inhibitor.
7. Any medical, geographic, or social factor making study participation impractical or precluding 1 month follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
MACE OR Myocardial Blush Grade 0/1 OR Distal Embolization OR Failure to Achieve ≥50% ST-segment Resolution | 30 days post-randomization
  The primary efficacy variable is the binary composite outcome with the following components:
  * The occurrence of any of the MACE outcomes (cardiovascular death, myocardial re-infarction, cardiogenic shock and new onset heart failure) at 30 days post-randomization.
  * Post-procedural Myocardial Blush Grade of either 0 (Failure of dye to enter the microvasculature or persistent "staining", suggesting leakage of the contrast medium into the extravascular space) or 1 (Dye enters slowly but fails to exit the microvasculature. Dye is present in the next injection (30 seconds)).
  * Post-procedural Distal embolization, defined as distal filling defect with an abrupt 'cut-off' in one of the peripheral coronary branches of the infarct related artery, distal to the angioplasty site following PCI).
  * Failure to achieve ≥50% ST-segment resolution post-procedure.

SECONDARY OUTCOMES:
Complete ST-segment Resolution. | 30 minutes
  Complete (≥70%) ST-segment resolution (worst lead) at 30 minutes post-PCI
CV Death, MI, Cardiogenic Shock or New Onset HF | 30 Days
  Composite of cardiovascular death, myocardial re-infarction, cardiogenic shock or new onset heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shamir Mehta, MD, Principal Investigator — McMaster University, Hamilton Health Sciences, Population Health Research Institute
Locations (3):
- Canada (3):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta - Mazankowski Alberta Heart Insitute, Edmonton, Alberta
  - Hamilton General Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta SR, Pinilla-Echeverri N, Tiong D, Kovalova T, Sheth T, Natarajan MK, Sibbald M, Velianou JL, Welsh R, Har B, Jolly SS, Valettas N, Schwalm JD, Tsang M, Khatun R, Mian R, Cunningham J, Ly E, McCready T, Bainey KR. Intracoronary Low-Dose Recombinant Tissue Plasminogen Activator in Primary PCI for ST-Segment Elevation Myocardial Infarction and Large Thrombus Burden: A Randomized Trial. J Am Coll Cardiol. 2026 Jan 27;87(3):238-248. doi: 10.1016/j.jacc.2025.10.008. Epub 2025 Oct 28. PMID 41194755